CLINICAL TRIAL: NCT06415123
Title: A Prospective, Randomized, Multi-center Study to Assess the Performance of MagnEtOs Flex Matrix Compared to Cellular Allograft in Patients Undergoing up to Four-level Instrumented poSterolatEral Lumbar/Thoraco-lumbar Fusion (PLF)
Brief Title: Study to Assess the Performance of MagnEtOs Flex Matrix Compared to Cellular Allograft
Status: Enrolling by invitation | Type: Observational
Sponsor: Research Source (Network)
Responsible Party: Sponsor
Other Study IDs: CT-003
Record Dates: First submitted 2024-05-09; First posted 2024-05-16 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Degenerative Disc Disease
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: MagnetOs Flex Matrix — MagnetOsTM Flex Matrix is a resorbable and osteoconductive bone graft for the repair of bony defects.

SUMMARY:
The purpose of this study is to demonstrate the performance of MagnetOs Flex Matrix in patients with leg pain and/or back pain.

DETAILED DESCRIPTION:
This is a prospective, randomized, multi-center study that intends to demonstrate the performance of MagnetOs Flex Matrix compared to Cellular Allograft in patients with leg pain and/or back pain requiring up to four-level instrumented PLF surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is able to read/be read, understand, and provide written informed consent and has signed the IRB approved informed consent.
2. Male or female patient ≥ 18 years old.
3. Patients with leg pain, and/or back pain requiring up to four-level instrumented posterolateral lumbar/thoraco-lumbar fusion (T11 - S1).
4. Failed conservative treatment (physical therapy, bed rest, medications, spinal injections, manipulations, or transcutaneous electrical nerve stimulation) for a minimum period of 3 months prior to study enrollment.

Exclusion Criteria:

1. Requires greater than four-level fusion or expected to need secondary intervention within one year following surgery.
2. Had prior PLF fusion or attempted PLF fusion at the involved levels.
3. Had previous decompression at the involved levels.
4. Women who are or intend to become pregnant within the next 12 months.
5. To treat conditions in which general bone grafting is not advisable.
6. In conditions where the surgical site may be subjected to excessive impact or stresses, including those beyond the load strength of fixation hardware (e.g., defect site stabilization is not possible).
7. In case of significant vascular impairment proximal to the graft site.
8. In case of severe metabolic or systemic bone disorders (e.g., osteogenesis imperfecta or Paget's Disease) that affect bone or wound healing.
9. In case of acute and chronic infections in the operated area (soft tissue infections; inflammation, bacterial bone diseases; osteomyelitis).
10. When intraoperative soft tissue coverage is not planned or possible.
11. Undergoing any procedure that allows MagnetOs to come in direct contact with the articular space.
12. Receiving treatment with medication interfering with calcium metabolism.
13. Has leg pain, and/or back pain related to benign or malignant tumor.
14. Has history or presence of active malignancy.
15. Has known substance abuse, psychiatric disorder, or a condition which, in the opinion of the investigator, may influence the healing or ability to comply with protocol requirements.
16. Is involved in active litigation relating to his/her spinal condition.
17. Has participated in an investigational study within 30 days prior to surgery for study devices

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient with leg pain and/or back pain requiring treatment with up to four-level instrumented posterolateral lumbar/thoraco-lumbar fusion (PLF) and who meet the following inclusion criteria and none of the exclusion criteria will be enrolled in the study. A patient is considered enrolled upon placement of the MagnetOs Flex Matrix during the surgical procedure. If the surgeon decides intra-operatively not to utilize the MagnetOs Flex Matrix, the patient will be considered a screen failure.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-06-11 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Posterolateral side fusion | 12 months post surgery
  The percentage of the posterolateral sides with bridging bone for the MagnetOs Flex Matrix and control treatments using CT-scans and determined by evidence of bridging trabeculae or continuous bony connection between superior and inferior transverse processes.

SECONDARY OUTCOMES:
Posterolateral lumbar/thoraco-lumbar fusion | 6 months post surgery
  Posterolateral lumbar/thoraco-lumbar fusion at Month 6 post-surgery assessed by CT-scans
Clinical outcome via Oswestry Low Back Pain Disability Questionnaire (ODI) | 12 months post-surgery
  Standard of care patient reported Oswestry Low Back Pain Disability Questionnaire (ODI) will be used to evaluate patient pain. On a scale of 0 to 6 with a score of 0 being no pain and a score of 5 being worst pain. A low score means a better clinical outcome. A high score means a worse clinical outcome.
Secondary Surgical Interventions (SSI's) | 12 months post-surgery
  Number of patients with revisions, re-operations, removals, supplemental fixations, and any other procedure that adjust or in any way remove part of the original implant configuration with or without replacement of the components within 12 months post-surgery. A low score (numbers of revisions, reoperations, etc.) means better safety outcome. A high score (numbers of revisions, reoperations, etc.) means a worse safety outcome.
Clinical outcome via neck visual analog scale (VAS) | 12 months post-surgery
  Standard of care patient reported neck visual analog scale (VAS) will be used to evaluate patient pain. On a scale of 0 to 10 with a score of 0 being no pain and a score of 10 being worst pain. A low score means a better clinical outcome. A high score means a worse clinical outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Michigan Orthopaedic Surgeons, Southfield, Michigan, United States

IPD SHARING:
Plan to Share IPD: No